CLINICAL TRIAL: NCT01441219
Title: Evaluation the Performance of Given Diagnostic System in Detection of Bleeding Events in the Small Bowel: a Single-arm Prospective Cohort Study.
Brief Title: Evaluation the Performance of Given Diagnostic System in Detection of Bleeding Events in the Small Bowel
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Results were obtained in another project.
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C2 in SB
Record Dates: First submitted 2011-08-02; First posted 2011-09-27 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Gastrointestinal Hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colon 2 (Experimental): using Colon 2 capsule in detecting bleeding events in small bowel
  Interventions: Device: Colon 2

INTERVENTIONS:
Device: Colon 2 — Ingest one colon 2 capsule
  Other Names: C2

SUMMARY:
Obscure gastrointestinal bleeding (OGIB) has been one of the most challenging area in the field of gastroenterology, as small bowel is beyond the reach of ordinary endoscopes like oesophagogastroduodenoscopy (OGD) and colonoscopy. Thanks for the latest technological advancement for investigating small intestine, we are now capable of obtaining intraluminal images safely through capsule endoscopy (CE). Its role in obscure gastrointestinal bleeding, Crohn's disease and other small bowel pathologies has already been proven, and nowadays it is suggested by various authorities to be the first-line modality among all small bowel investigations.

The investigators group has showed that CE can alter the clinical management of patients with OGIB - patients with negative CE has lower rebleeding rate, and therefore we may adopt a conservative approach for them. Although supported by some other group as well, conflicting results were still reported in the literature about the out-come of these patients. The main criticisms for these studies are that, CE can only identify 61% of the underlying small bowel bleeding pathology, and one can never ascertain the outcome of patients with negative CE examination. Apparently there is still room for improvement in the current CE technology.

DETAILED DESCRIPTION:
Newer generation of CE (PillCam ColonTM) has been developed to investigate the large bowel. It is different from small bowel CE that it consists of two cameras at both ends of the capsule, so as to enhance the coverage of colonic mucosa visualization. An improved generation of this colon capsule, named PillCam Colon 2TM, is also in its developmental phase. With the new "adaptive frame rate" (AFR) technology, the CE optimizes the visual coverage of the bowel by increasing the frame rate up to 35 frames per second when the capsule is moving quickly in certain areas, while decreasing the frame rate down to 4 frames per second when the capsule is moving slowly or remains stationary so as to conserve the battery life. Preliminary data from colorectal cancer screening has shown that it could improve the diagnostic yield of colonic polyps.

The investigators hypothesize that, by re-programming the PillCam Colon 2TM so as to initiate AFR since ingestion, it could improve the visualization of small intestinal lumen and hence improves the sensitivity of small bowel CE examination.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with overt GI bleeding (hematemesis, coffee-grounds, rectal bleeding and/or melena) with negative OGD but not critically ill, who should read positive on small bowel investigation (SBI)
2. Patients with occult GI bleeding (Faecal occult blood test,FOBT +)
3. Patients with suspected arteriovenous(AV) malformations.
4. Patients treated with nonsteroidal antiinflammatory drugs (NSAIDs)
5. Patients with active Crohn's disease(CD), with no evidence of obstruction

Exclusion Criteria:

1. In patients with known or suspected gastrointestinal obstruction, strictures, or fistulas based on the clinical picture or pre-ingestion testing and profile.
2. In patients with cardiac pacemakers or other implanted electromedical devices.
3. In patients with dysphagia or other swallowing disorders.
4. Unable to obtain informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield for bleeding events in the small bowel | 1 year
  Review the capsule video to detect the bleeding events.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph JY Sung, MD, Principal Investigator — CUHK
Locations (1):
- Prince of Wales Hospital, Hong Kong, China